CLINICAL TRIAL: NCT02304614
Title: The Use of 3D Surface Imaging in the Objective Assessment of Breast Conserving Therapy
Acronym: 3DBCT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR4252
Record Dates: First submitted 2014-11-27; First posted 2014-12-02 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Patients who have undergone Breast conserving Therapy
  Interventions: Other: 3D surface imaging using a non portable and portable camera; Other: Patient reported outcome measure (PROM): BREAST-Q; Other: 2D photography; Other: Applanation Tonometry

INTERVENTIONS:
Other: 3D surface imaging using a non portable and portable camera — The participant will have 3D surface imaging taken of their breasts (the face will not be shown)
  Other Names: 3D photography
Other: Patient reported outcome measure (PROM): BREAST-Q — The participant will answer the BREAST-Q questionnaire. This is a patient reported outcome measurement of satisfaction and quality of life after BCT
Other: 2D photography — The participant will have standard medical photography of their breasts (the face will not be shown)
  Other Names: medical photography
Other: Applanation Tonometry — A small 300g disc is placed on the breast to measure the surface area of contact with the breast to measure compressibility
  Other Names: Measurement of breast compressibility

SUMMARY:
3D surface imaging has been used in the objective evaluation of cosmetic outcome of oncoplastic procedures such as breast reconstruction and lipofilling, however there is only one article published relating to Breast Conserving Therapy (BCT).

The aim of this study is to assess the use 3D surface imaging as a tool in the assessment of symmetry of outcome following breast conserving therapy. The results of the surface imaging will be correlated with patient satisfaction, using the BREAST-Q, which is a validated patient questionnaire and correlated with panel assessment by an independent panel of two surgeons, one clinical oncologist and one breast care nurse.

DETAILED DESCRIPTION:
BCT is the most common breast surgical oncological procedure performed with approximately 28,500 patients undergoing this operation every year. In breast cancer surgery, the primary aim of removing the cancer must be reconciled with the secondary aim of preserving breast aesthetics. Objective analysis of cosmetic outcome measures in breast surgery has been lacking, however 3D surface imaging is beginning to show promise in this area. Having a robust tool for objective assessment of outcomes may facilitate critical appraisal of techniques and therefore surgeon learning.

Currently the cosmetic success of an operation can be subjectively evaluated by patients' and surgeons' visual assessment. Patient reported outcome measures (PROMs) are instruments to measure any aspect of a patient's health status. Various PROMs have been used to evaluate patients' satisfaction after breast cancer treatment. For example, the BREAST-Q was developed quantitatively and qualitatively to measure patients' perceptions before and after breast reconstruction by examining quality of life domains (psychosocial well-being, physical well-being, sexual well-being) and satisfaction domains (satisfaction with breasts, satisfaction with outcome, satisfaction with care). When using any of these PROMs, accuracy and reproducibility are not measurable; the results are the subjective views of the patient. While the patient opinion of her own appearance is clearly the most important outcome after local oncological control, for the purposes of objective comparison between groups of patients, surgeons and over time, independent clinicians (and / or lay people) may be recruited to perform a 'panel assessment' of photographs in which the various aspects of cosmesis such as breast shape, size and cleavage are considered in addition to overall appearance. However such assessments are still subjective and often lack accuracy and reproducibility.

There have been many attempts to derive objective measures of outcome. In the 1970's, Edstron et al described 'split and reversed negatives' where photographic negatives of the left and right breast were made and laid next to the non-negative right and left breast. The constructed images of perfectly symmetrical breasts were compared with the original photographs of the patients' breasts. More recently two software systems have been developed to objectively evaluate the aesthetic surgical outcomes of breast surgery using 2D photographs. The Breast Analyzing Tool (BAT©) evaluates symmetry by comparing breast area, breast circumference and nipple position between the breasts. The Breast Cancer Conservative Treatment cosmetic result (BCCT.core) also analyses colour differences and the scar appearance in addition to asymmetry calculations.

The use of 3D surface imaging in the clinical setting was first described by Burke and Beard in 1967 to analyze facial structures. Over the last fifteen years 3D imaging has been used as a research and clinical tool in aesthetic, oncoplastic and reconstructive breast surgery. Initial studies established optimal technique to obtain images and tested accuracy and reproducibility. 3D imaging is currently used to simulate for the patient what a cosmetic augmentation might achieve in terms of size and shape. It has been demonstrated that simulated images are accurate and patients felt they helped them to choose the implant.

In terms of oncoplastic reconstructive surgery 3D surface imaging has been used in the objective evaluation of cosmetic outcome of oncoplastic procedures such as breast reconstruction and lipofilling, however there is only one article published relating to Breast Conserving Therapy (BCT). Moyer et al analyzed twenty three patients who had undergone BCT and compared volume and asymmetry. They found that there was a positive correlation between percentage of breast parenchyma excised and asymmetry. The location of the cancer, age of the patient and need for multiple operations did not influence cosmetic results but the sample size was small and therefore likely underpowered.

The aim of this study is to assess the use 3D surface imaging as a tool in the assessment of symmetry of outcome following breast conserving therapy. The results of the surface imaging will be correlated with patient satisfaction, using the BREAST-Q, which is a validated patient questionnaire and correlated with panel assessment by an independent panel of two surgeons, one clinical oncologist and one breast care nurse.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* No age limit
* underwent unilateral breast conserving surgery at The Royal Marsden NHS Foundation Trust (RMH)
* underwent adjuvant whole breast radiotherapy at RMH
* attending for their annual surveillance mammogram
* between one and five and half years after surgery (rounded to nearest whole year)

Exclusion Criteria:

* undergone surgery to the contralateral breast (breast conserving surgery, symmetrisation or mastectomy)
* undergone further surgery to the affected breast subsequent to BCT (eg lipofilling or other reconstruction).
* unable to stand for long enough to have clinical photos (approximately 10 minutes)
* unable to answer the BREAST-Q questionaire (e.g. learning difficulties)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have undergone Breast Conserving Therapy at least one year ago
Sampling Method: Non-Probability Sample
Enrollment: 346 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2017-03-22 (Actual); Study Completion 2020-12-24 (Estimated)

PRIMARY OUTCOMES:
A multivariate model using clinical risk factors to predict percentage volume asymmetry | measured on day of imaging

SECONDARY OUTCOMES:
Comparison of panel assessment of the symmetry of outcome of BCT by independent clinicians using 2D and 3D photography with patient reported outcome using satisfaction with breasts domain of the breast conservation module of the BREAST-Q | measured on day of imaging
Establishment of the most reproducible method to measure focal deficits using 3D surface imaging | measured on day of imaging
Comparison of the volume measurements in women who have undergone BCT as measured by VECTRA XT (non portable 3D surface imaging device) and VECTRA H1 (portable 3D surface imaging device) | measured on day of imaging
Comparison of compressibility of treated and untreated breasts as measured by applanation tonometry | measured on day of imaging

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E Rusby, DM FRCS, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, United Kingdom